CLINICAL TRIAL: NCT06671119
Title: REvision of VSG with Ablation of the Mucosa Procedure
Acronym: REVAMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Christopher McGowan (Other)
Responsible Party: Sponsor-Investigator, Dr. Christopher McGowan, Co-Founder/Co-CEO/Chief Medical Officer, True You Weight Loss
Organization: True You Weight Loss (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20242649
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Obesity and Obesity-related Medical Conditions; Obesity and Overweight; Obesity Prevention; Obesity Recidivism
Keywords: obesity; obesity and overweight; endoscopic bariatric therapy; ablation; gastric mucosal ablation; GMA
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Gastric Mucosal Ablation (GMA) following sleeve gastrectomy (Experimental): Subjects will undergo endoscopic Gastric Mucosal Ablation (GMA) following sleeve gastrectomy. This will be performed by an experienced endoscopist specialized in bariatric endoscopy in a single endoscopic session.
  Interventions: Device: Gastric Mucosal Ablation (GMA)

INTERVENTIONS:
Device: Gastric Mucosal Ablation (GMA) — Endoscopic Gastric Mucosal Ablation (GMA) after sleeve gastrectomy

SUMMARY:
The purpose of this study is to evaluate the feasibility, safety, and tolerability of endoscopic selective gastric mucosal ablation (GMA) using argon plasma coagulation after sleeve gastrectomy. In this study, GMA will be performed on patients who have experienced weight regain following an initial successful response to sleeve gastrectomy.

DETAILED DESCRIPTION:
Obesity is a multifaceted chronic disease associated with substantial morbidity and mortality, leading to conditions like diabetes, cardiovascular diseases, and malignancies. Bariatric procedures, such as the sleeve gastrectomy, stand out as the current most effective long-term treatments for obesity. Despite its effectiveness, a significant number of patients experience weight regain during long-term follow-up. Endoscopic minimally invasive bariatric intervention has been proposed as a viable, safe, and effective option for the treatment of weight regain after SG. Gastric mucosal ablation (GMA), in particular, is hypothesized to be a safe and effective endoscopic revisional treatment for weight regain following sleeve gastrectomy based on previous positive pre-clinical and clinical studies. To investigate the feasibility, safety, and tolerability of GMA after sleeve gastrectomy, a single procedure is designed to ablate the gastric mucosa of the pseudo greater curvature created after the sleeve gastrectomy in a single endoscopic session. We hypothesize that endoscopic selective ablation of the gastric mucosa after sleeve gastrectomy is effective as a revisional treatment for weight regain and will result in significant metabolic improvements.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients who have:

   1. BMI of 30 kg/m2 or greater, AND
   2. regained at least 25% of the total weight lost after initial successful response to sleeve gastrectomy. defined as Excess Weight Loss (EWL) greater than 50% or Total Body Weight Loss (TBWL) exceeding 20%
2. Must have undergone SG at least three years before the time of enrollment
3. Age range: 22 - 60 years
4. Must agree to refrain from using weight loss medications such as Meridia, Saxenda, Januvia, Xenical, Duromine, GLP-1 agonists (e.g., Ozempic, Wegovy) and dual GLP-1/GIP agonists (e.g., Mounjaro, Zepbound), as well as any over-the-counter weight loss medications or supplements throughout the study.
5. Women of childbearing potential (WOCBP) must agree to use acceptable contraception methods.
6. Must agree not to donate blood during participation in the study.
7. Should be able to comply with study requirements, understand, and sign the Informed Consent Form.
8. Stable weight defined as a fluctuation of less than 5% for at least 3 months prior to the screening visit.
9. Should have a history of failure to lose weight using conventional diet and lifestyle therapies.
10. Must have reliable access to wifi and/or internet services.
11. Must express willingness to comply with the substantial lifelong dietary restrictions required by the procedure.

Exclusion Criteria:

1. Inadequate response to sleeve gastrectomy
2. Patients requiring exogenous insulin.
3. HbA1c > 8.5%
4. Pregnant or breast-feeding or intending to get pregnant during the study.
5. Unwilling or unable to complete the Visual Analogue Scale for pain assessment, patient questionnaires, or comply with study visits and other study procedures as required per protocol.
6. History of diabetic ketoacidosis or hyperosmolar nonketotic coma.
7. Previous use of any types of insulin for > 1 month (at any time, except for treatment of gestational diabetes).
8. Change in diabetic treatment within the last three months.
9. Use of glucose-lowering drugs for diabetes mellitus treatment with the exception of sulfonylurea (SU), biguanides and sodium-dependent glucose co-transporter 2 (SGLT-2) inhibitors.
10. GLP-1 use in the preceding 6 months.
11. Known autoimmune disease, other than autoimmune thyroid disease, which is adequately replaced, including but not limited to celiac disease, or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder.
12. Previous endoscopic bariatric procedures or conditions, prior intra-gastric balloon or another gastric implant.
13. History of diabetic gastroparesis.
14. Known active hepatitis or active liver disease other than Non-Alcoholic Fatty Liver Disease or Non-Alcoholic Steatohepatitis.
15. Acute gastrointestinal illness in the previous 7 days.
16. Known history of irritable bowel syndrome, radiation enteritis, or other inflammatory bowel disease, such as Crohn's disease.
17. Known history of a structural or functional disorder of the esophagus that may impede passage of the device through the gastrointestinal tract or increase the risk of esophageal damage during an endoscopic procedure, including Barrett's esophagus, esophagitis, dysphagia, achalasia, stricture/stenosis, esophageal varices, esophageal diverticula, esophageal perforation, or any other disorder of the esophagus.
18. Known history of a structural or functional disorder of the esophagus, including any swallowing disorder, esophageal chest pain disorders, or drug-refractory esophageal reflux symptoms.
19. Known history of a structural or functional disorder of the stomach, including gastroparesis, gastric ulcer, chronic gastritis, gastric varices, hiatal hernia (>3 cm), cancer, or any other disorder of the stomach.
20. Known history of chronic symptoms suggestive of a structural or functional disorder of the stomach, including any symptoms of chronic upper abdominal pain, chronic nausea, chronic vomiting, chronic dyspepsia, or symptoms suggestive of gastroparesis, including post-prandial fullness or pain, post-prandial nausea or vomiting, or early satiety.
21. Currently have ongoing symptoms suggestive of intermittent small bowel obstruction, such as recurrent bouts of post-prandial abdominal pain, nausea, or vomiting.
22. Active H. pylori infection (Subjects with active H. pylori may continue with the screening process if they are treated with an appropriate antibiotic regimen, and eradication has been confirmed).
23. History of coagulopathy, upper gastrointestinal bleeding conditions such as ulcers, gastric varices, strictures, congenital or acquired intestinal telangiectasia.
24. Current use of anticoagulation therapy.
25. Obligate use of anti-inflammatory drugs that cannot be suspended for a minimum of 4 weeks post procedure.
26. Use of systemic glucocorticoids (excluding topical or ophthalmic application or inhaled forms) for more than 10 consecutive days within 90 days prior to the Screening Visit.
27. Use of drugs known to affect GI motility (e.g., Metoclopramide).
28. Receiving any weight loss medications such as Meridia, Xenical, Saxenda, Januvia, Duromine, GLP-1 agonists, GIP/GLP-1 dual agonists, or over-the-counter weight loss medications at screening.
29. Untreated/inadequately treated hypothyroidism, defined as an elevated Thyroid-Stimulating Hormone (TSH) level at Screening; if on thyroid hormone replacement therapy, must be on a stable dose for at least 6 weeks prior to Screening.
30. Persistent Anemia, defined as Hemoglobin <10 g/dL.
31. Significant cardiovascular disease including a known history of valvular disease, or myocardial infarction, heart failure, transient ischemic attack, or stroke within the last 6 months.
32. Known moderate or severe chronic kidney disease (CKD), with estimated glomerular filtration rate (eGFR) <45 ml/min/1.73m2 (estimated by MDRD).
33. Known immunocompromised status, including but not limited to individuals who have undergone organ transplantation, chemotherapy, or radiotherapy within the past 12 months, who have clinically significant leukopenia, who are positive for the human immunodeficiency virus (HIV) or whose immune status makes the subject a poor candidate for clinical trial participation in the opinion of the Investigator.
34. Active systemic infection.
35. Known active malignancy within the last 5 years (with the exception of treated basal cell or treated squamous cell carcinoma).
36. Subjects with an established diagnosis of Multiple Endocrine Neoplasia syndrome type 1.
37. Not a candidate for surgery or general anesthesia.
38. Active illicit substance abuse or alcoholism.
39. Current smoker or smoking history in the last six months.
40. Participating in another ongoing clinical trial of an investigational drug or device.
41. Any other mental or physical condition which, in the opinion of the Investigator, makes the subject a poor candidate for clinical trial participation.
42. Other medical conditions that do not allow for an endoscopic procedure.

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Total Body Weight Loss (TBWL) from Baseline | 6 Months
  Measure percent change in total body weight over time following endoscopic GMA. TBWL = pre-op weight - post op body weight. % TBWL is the fraction of body weight expressed in percentage term

SECONDARY OUTCOMES:
Rate of Safety Complications according to Clavien-Dindo Classification | Month 1, Month 2, Month 3, Month 4, Month 6, Month 7, Month 8, Month 9, Month 10, Month 11, Month 12
  Occurrence of complications according to the Clavien-Dindo classification
Rate of Adverse Events (AE) | Month 1, Month 2, Month 3, Month 4, Month 6, Month 7, Month 8, Month 9, Month 10, Month 11, Month 12
  Occurrence of Adverse Events along with AE Type, severity, and relationship to treatment.
Post-operative Pain Assessment | Month 1, Month 2, Month 3, Month 4, Month 6, Month 7, Month 8, Month 9, Month 10, Month 11, Month 12
  Visual Analog Scale pain score at baseline compared to postoperative follow-up visits. The VAS Pain Scores range from 0 (minimum) to 10 (maximum), where 0 represents no pain and 10 represents the maximum level of pain, with higher scores indicating greater intensity of postoperative pain.
Percent Change in Total Body Weight Loss (TBWL) from Baseline | Month 12
  Measure percent change in total body weight over time following endoscopic GMA. TBWL = pre-op weight - post op body weight. % TBWL is the fraction of body weight expressed in percentage term
Quality of Life Assessment | 6 Months
  Baseline quality of life assessment scores compared to 6 Month quality of life assessment scores. Quality of life score assessed and measured by the 36-Item Short Form Survey and The Impact of Weight on Quality of Life-Lite questionnaires. Scoring for both questionnaires range from 0 (minimum) to 100 (maximum). Higher scores for both questionnaires indicate higher quality of life.
Glucose Homeostasis Assessment | 3 Months, 6 Months
  Baseline measured fasting glucose, HOMA-IR, and HbA1c levels compared to post-intervention fasting levels at 3 Months and 6 Months using laboratory testing.
Serum Levels of Lipids Assessment | 3 Months, 6 Months
  Baseline compared to post-intervention fasting serum lipids levels at 3 Months and 6 Months measured by laboratory testing.
Gastric Sensory Function Assessment | 3 Months, 6 Months
  Volume to comfortable fullness and Maximum Tolerated Volume measured using a visual analog scale at 3 Months and 6 Months. Volume to Comfortable Fullness and Maximum Tolerated Volume scores both range from 0 (minimum) to 100 (maximum) with a lower score indicating a smaller required volume to reach comfortable fullness and maximum fullness.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher McGowan, MD, MSCR, Principal Investigator — True You Weight Loss
Locations (1):
- True You Weight Loss, Cary, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bulajic M, Vadala di Prampero SF, Boskoski I, Costamagna G. Endoscopic therapy of weight regain after bariatric surgery. World J Gastrointest Surg. 2021 Dec 27;13(12):1584-1596. doi: 10.4240/wjgs.v13.i12.1584. PMID 35070065
- [Background] Lauti M, Kularatna M, Hill AG, MacCormick AD. Weight Regain Following Sleeve Gastrectomy-a Systematic Review. Obes Surg. 2016 Jun;26(6):1326-34. doi: 10.1007/s11695-016-2152-x. PMID 27048439